CLINICAL TRIAL: NCT05854342
Title: Evaluation of the Effects of Bicarbonate-calcium Water in Premenopausal and Postmenopausal Women as a Prevention of Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salerno (Other)
Collaborators: San Giuseppe Moscati Hospital (Other)
Responsible Party: Principal Investigator, Luca Rastrelli, Principal Investigator Full Professor Luca Rastrelli, University of Salerno
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CECN/1522
Record Dates: First submitted 2023-03-14; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Osteoporosis Risk
Keywords: bicarbonate-calcium water

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bicarbonate-calcium water (Experimental): participants of this group drink bicarbonate-calcium water
  Interventions: Other: bicarbonate-calcium water
- low mineral water (No Intervention): participants of this group drink low mineral water

INTERVENTIONS:
Other: bicarbonate-calcium water — water with high content of bicarbonate and calcium, low sodium
  Arms: bicarbonate-calcium water

SUMMARY:
The goal of this clinical trial is to evaluate the effect of bicarbonate-calcium water for the prevention of osteoporosis. Participants are women in pre- or post- menopausal state. The intervention group must drink bicarbonate-calcium water while the control group low mineral water

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged ≥40 years
* Menopausal women, period of early menopause 1-10 years

Exclusion Criteria:

* Inclusion in other study protocols
* estrogen-replacement hormone therapy
* osteoporosis therapy
* corticosteroid therapy
* insulin therapy.
* calcium supplementation
* kidney diseases of medium-severe level
* liver diseases of medium-severe level
* severe osteoporosis

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
calcium (mg/dL) | 0-3-6 month
  change of some physiological parameters concentration related to calcium metabolism measured by blood laboratory tests
25-OH vitamin D (ng/mL) | 0-3-6 month
  change of physiological parameter concentration related to calcium metabolism
osteocalcin (ng/mL) | 0-3-6 month
  change of physiological parameter concentration related to calcium metabolism
Parathyroid hormone (pg/mL) | 0-3-6 month
  change of physiological parameter concentration related to calcium metabolism

SECONDARY OUTCOMES:
NMR metabolomic profile and applications of Metabolomics in calcium metabolism | 0-3-6 month
  Metabolomic profile of serum related to calcium metabolism by NMR proton Nuclear Magnetic Resonance spectroscopy (1H-NMR) Metabolomics aims at the quantitative analysis of all metabolites in a biological system, as well as their composition, interactions, and responses to interventions or a specific physiological state. The metabolomics approach correlates broad biochemical changes with health and disease states, and advanced statistical metabolic modeling allows the identification of biomarkers, enabling the quantification of low-molecular-weight metabolites

OTHER OUTCOMES:
changes cholesterol total (mg/dL) | 0-3-6 month
  change of physiological parameter concentration related to lipidic profile measured by blood laboratory tests
changes cholesterol HDL (mg/dL) | 0-3-6 month
  change of physiological parameter concentration related to lipidic profile measured by blood laboratory tests
changes cholesterol LDL (mg/dL) | 0-3-6 month
  change of physiological parameter concentration related to lipidic profile measured by blood laboratory tests
changes glycemia (mg/dL) | 0-3-6 month
  change of physiological parameter concentration related to glycemic profile measured by blood laboratory tests

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salerno, Salerno, Italy

REFERENCES:
- [Background] Meunier PJ, Jenvrin C, Munoz F, de la Gueronniere V, Garnero P, Menz M. Consumption of a high calcium mineral water lowers biochemical indices of bone remodeling in postmenopausal women with low calcium intake. Osteoporos Int. 2005 Oct;16(10):1203-9. doi: 10.1007/s00198-004-1828-6. Epub 2005 Mar 3. PMID 15744450
- [Background] Wynn E, Krieg MA, Aeschlimann JM, Burckhardt P. Alkaline mineral water lowers bone resorption even in calcium sufficiency: alkaline mineral water and bone metabolism. Bone. 2009 Jan;44(1):120-4. doi: 10.1016/j.bone.2008.09.007. Epub 2008 Sep 26. PMID 18926940

DOCUMENTS (3):
  • Study Protocol (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT05854342/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT05854342/SAP_001.pdf
  • Informed Consent Form (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT05854342/ICF_002.pdf